CLINICAL TRIAL: NCT04057443
Title: Impact of a Nutritional and Physical Exercise Intervention Program on Oncological Treatment Completion in Patients ≥70 Years Old With Malignant Hemopathies:ICOSENIORHEM Randomized Clinical Trial
Brief Title: Nutritional and Physical Exercise Intervention in Older Patients With Malignant Hemopathies
Acronym: ICOSENIORHEM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maite Antonio, MD, Phd (Other)
Collaborators: Institut d'Investigació Biomèdica de Bellvitge (Other); University of Barcelona (Other); Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor-Investigator, Maite Antonio, MD, Phd, Coordinator Oncohematogeriatrics Unit. Institut Català d'Oncologia, L'Hospitalet de Llobregat
Organization: L'Hospitalet de Llobregat (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ICOSENIORHEM; PR157/18 (Other: Independent review board)
Record Dates: First submitted 2019-06-11; First posted 2019-08-15 (Actual); Last update posted 2019-08-30 (Actual); Status verified 2019-08

CONDITIONS: Hematologic Malignancy; Old Age; Debility
Keywords: older; physical exercise; nutrition support; hematologic malignancies; geriatric assessment; geriatric intervention
MeSH Terms: conditions — Hematologic Neoplasms; Frailty; Motor Activity | interventions — Nutritional Support; Exercise

STUDY DESIGN:
Intervention Model Description: Parallel design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Patients in the intervention group will follow the standard treatment and follow-uo according to the clinical protocol of the institution and will participate in an intervention program with physical exercise and nutritional support during the period in which they are receiving oncological treatment or for a maximum period of 6 months.
  Interventions: Other: Nutritional support; Other: Physical exercise; Drug: Hematologic Drug
- Control group (Active Comparator): The patients of the control group will follow the standard treatment and follow-up according to the clinical protocol of the institution.
  Interventions: Drug: Hematologic Drug

INTERVENTIONS:
Other: Nutritional support — Nutritional support will be given to all patients according with their nutritional body composition parameters (Nutritional assessment and sarcopenia evaluation). It could be diet counselling, oral supplemented nutrition, enteral nutrition o parenteral nutrition.
  Arms: Intervention group
Other: Physical exercise — The exercise program, designed, applied and monitored by research staff of the Physiology Unit, will have duration of 24 weeks (6 months). The program will have a mixed structure, the participants in an individual way fulfill their training and attend group sessions (8 subjects). In addition, 3 days a week should conduct sessions that will focus on the work of balance and general strength.
  Arms: Intervention group
Drug: Hematologic Drug — The patients of the control group will follow the standard treatment and follow-up according to the clinical protocol of the institution.

SUMMARY:
Clinical trial to analyze the impact of nutrition and physical exercise intervention program on the completion of treatment in older patients 70 years or older with malignant hemopathology

DETAILED DESCRIPTION:
OBJECTIVE:

This study aims to determine wether a geriatric intervention based on an individualized program of physical exercise and nutritional support improves the ability to complete oncological treatment at the doses and time initially planned in patients ≥ 70 years affected by hematological malignancies.

DESIGN:

Prospective, clinical trial, randomized, parallel and open groups.

SETTING:

Patients ≥ 70 years recently diagnosed of malignant hematological pathology in a comprehensive cancer center

INTERVENTION:

All those patients who meet the inclusion criteria and agree to participate, will sign the corresponding informed consent and will be assessed through a CGA (comprehensive geriatric assessment), that includes the performance of a physical condition test (SPPB), and randomized to the study group or control group. Patients in the study group will participate in an intervention program with nutritional support and physical exercise during the period in which they are receiving oncological treatment or for a maximum period of 6 months. The patients of the control group will pass to follow up. All patients, regardless of the branch of study to which they are assigned, will receive the oncological treatment indicated by their doctor and a standard follow-up according to the current care protocols in the center.

DETERMINATIONS:

Main variable: proportion of adherence to treatment calculated as the percentage between the dose administered and the prescribed. Adherence over 80% will be considered acceptable.

Secondary variables: geriatric, nutritional and physical-condition parameters before and after the intervention, quality of life before and after the intervention, toxicity and complications during treatment and response to treatment.

ELIGIBILITY:
Inclusion Criteria:

* hematological pathology (myelodysplastic syndromes, lymphoproliferative syndromes, multiple myeloma)
* considered able to practice physical exercise
* signed informed consent

Exclusion Criteria:

* other hematological pathology
* considered unable to practice physical exercise

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-04-11 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Adherence to oncological treatment | Change from baseline and after finishing treatment or 6 months
  Percentage between the dose administered and the prescribed.

SECONDARY OUTCOMES:
Risk of vulnerability | Baseline versus 6 months (end of intervention) versus 12 months
  Vulnerable Elders Survey (VES-13) (numeric variable)
Geriatric assessment | Baseline versus 6 months (end of intervention) versus 12 months
  Geriatric Assessment in Hematology (GAH scale) (numeric variable)
Nutritional screening | Baseline versus 6 months (end of intervention) versus 12 months
  Mini-Nutritional Assessment (MNA) (numeric variable)
Functional capacity | Baseline versus 6 months (end of intervention) versus 12 months
  Basic activities of daily life (ABVD) - (Barthel scale) and instrumental activities of daily life (IADL) (Lawton-Body scale), fatigue (Borg scale) (numeric variable)
Physical condition screening | Change from baseline versus 6 months (end of intervention) versus 12 months
  Short Portable Physical Performance (SPPB) test. Numeric variable.
Physical condition tests | Baseline versus 6 months (end of intervention) versus 12 months
  Walking test 4 metres, Up-and-go test (seconds)
Body mass index | Baseline versus 6 months (end of intervention) versus 12 months
  Weight and height will be combined to report body mass index (BMI) in kg/m2
Anthropometric evaluation | Baseline versus 6 months (end of intervention) versus 12 months
  Anthropometric evaluation of waist, hip, arm, thigh and leg perimeters (cm).
Body composition | Baseline versus 6 months (end of intervention) versus 12 months
  Body mass measured with electrical bioimpedance
Performance of muscular strength | Baseline versus 6 months (end of intervention) versus 12 months
  Strength measured by Isometric dynamometry of hands (hand grip) and legs (flex-extension) (KgF)
Functional capacity assessment | Change from baseline versus 6 months (end of intervention) versus 12 months
  6-minute walk test to assess functional capacity.
Assessment of lower limbs strengh | Change from baseline versus 6 months (end of intervention) versus 12 months
  Test to sit and get up in 30 seconds
Average number of exercise sessions completed | Through study completion, an average of 6 months
  Number of exercise sessions completed by each participant in the intervention group.
Incidence of adverse effects | Through study completion, an average of 6 months
  Frequency and severity of adverse effects according to CTCAE v4.
Quality of life Assessment | Change from baseline versus 6 months (end of intervention) versus 12 months
  Quality of Life Assessment: European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (QLQ)for old patients with cancer. (EORTC QLQ-ELD14): numeric variable.
Disease progression | Change from baseline and after 2 years
  Time to treatment failure, time to disease progression or death from any cause, and time to disease progression
Survival | Change from baseline and after 2 years
  Disease-free survival, overall survival, and cancer-specific survival.

CONTACTS AND LOCATIONS:
Overall Officials: Maite Antonio, MD,PhD, Principal Investigator — Institut Català d'Oncologia
Locations (1):
- Institut Català d'Oncologia, L'Hospitalet de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ernst M, Wagner C, Oeser A, Messer S, Wender A, Cryns N, Brockelmann PJ, Holtkamp U, Baumann FT, Wiskemann J, Monsef I, Scherer RW, Mishra SI, Skoetz N. Resistance training for fatigue in people with cancer. Cochrane Database Syst Rev. 2024 Nov 28;11(11):CD015518. doi: 10.1002/14651858.CD015518. PMID 39606939